CLINICAL TRIAL: NCT04341272
Title: Intermittent Pneumatic Compression of the Upper Extremity for Post-Operative VTE Prophylaxis: A Pilot Randomized Trial
Brief Title: Intermittent Pneumatic Compression of the Upper Extremity for Post-Operative VTE Prophylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Preeti R. John, MD, MPH, FACS, Clinical Assistant Professor, Baltimore VA Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HP-00051138
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Venous Thromboses
MeSH Terms: conditions — Venous Thrombosis | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upper Extremity Compression Device (Active Comparator): Patients randomized to have pneumatic compression device placed on upper extremity following surgery
  Interventions: Device: Intermittent Pneumatic Compression Device (FDA approved)
- Control (Other): Patients randomized to have pneumatic compression device placed on lower extremity following surgery
  Interventions: Device: Intermittent Pneumatic Compression Device (FDA approved)

INTERVENTIONS:
Device: Intermittent Pneumatic Compression Device (FDA approved) — Compression Device placed on either upper or lower extremity for DVT prophylaxis following surgery

SUMMARY:
Venous thromboembolism (VTE) is an important cause of morbidity and mortality following surgery.A combination of chemical and mechanical prophylaxis using lower extremity compression devices (CD) is recommended in patients who are considered at 'moderate risk' (Caprini score 2 - 4) or 'high risk' (Caprini score > 4) of developing VTE.

The aim of this study was to determine whether upper extremity (UE) CD are as effective as lower extremity (LE) CD in preventing VTE following surgery. A total of 106 patients were recruited.

DETAILED DESCRIPTION:
Hospitals throughout the United States currently utilize mechanical compression devices on patients' limbs for prevention of blood clots, in addition to blood thinning medication - heparin. The compression devices act by affect blood clotting mechanism and there is evidence from previous research studies that blood is less likely to develop clots when these compression devices are placed on the arms or legs.

The use of compression devices on arms and legs is within standard of care, but use on legs tends to be more common.

Research studies have shown that use of compression devices in combination with heparin is more effective in preventing blood clots than either one alone.

Not many clinicians remember the option of placing compression devices on arms, and patients who do not get compression devices placed on their legs following surgery, often get only medication (heparin) with no compression device placed at all.

This study will compare the effectiveness of compression devices used on patients' arms with those used on patients' legs, at preventing blood clots. Non-invasive ultrasound studies will be used after surgery to check for blood clots in the legs.

ELIGIBILITY:
Inclusion Criteria:

• Males aged > 18 years who could provide informed consent

Exclusion Criteria:

* Patients on coumadin or post-operative therapeutic heparin
* Known history of venous thromboembolism (VTE)
* Known history of hematological disorders
* Diagnosed malignancy requiring or undergoing treatment
* Presence of upper extremity arterio-venous access for hemodialysis
* Females were excluded to eliminate the confounding thrombogenic effect of estrogen.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
venous thromboembolic event following surgery | within 45 days following surgery
  venous thrombosis (VT) or pulmonary embolism (PE): number of screening lower extremity venous duplex ultrasound studies showing VT and any CT scans showing PE in symptomatic patients

CONTACTS AND LOCATIONS:
Overall Officials: Preeti R John, MD, MPH, FACS, Principal Investigator — Baltimore VA Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Priliminary data published in Journal of American College of Surgeons abstract — https://www.journalacs.org/article/S1072-7515(16)31034-1/abstract